CLINICAL TRIAL: NCT05034939
Title: FLEX Vessel Prep Prior to the Treatment of Obstructive Lesions in the Native Arteriovenous Dialysis Fistulae
Brief Title: FLEX Vessel Prep Prior to Angioplasty in Native Arteriovenous Fistulae (AVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMG-2021-001
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Arteriovenous Fistula Stenosis
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FLEX Vessel Prep System followed with PTA (TEST arm) (Active Comparator): FLEX Vessel Prep System is used to create circumferential, continuous micro-incisions along the length of the stenosis by performing a retrograde pullback through the lesion. Following FLEX, standard balloon angioplasty is performed with an uncoated PTA balloon sized to meet the reference vessel diameter, according to its corresponding instructions for use. Once advanced to the lesion, the balloon should be inflated according to the site's standard of care.
  Interventions: Device: FLEX Vessel Prep System
- PTA only (CONTROL arm) (Active Comparator): Standard Balloon angioplasty is performed with an uncoated PTA balloon sized to meet the reference vessel diameter, according to its corresponding instructions for use. Once advanced to the lesion, the balloon should be inflated according to the site's standard of care.
  Interventions: Device: Angioplasty

INTERVENTIONS:
Device: FLEX Vessel Prep System — The FLEX Vessel Prep System™ is an over-the-wire sheathed catheter with a three-strut treatment element near the distal tip. As the device is pulled back in a retrograde fashion through the target lesion, the Treatment Element "flexes" providing continuous engagement along the lesion to create controlled depth micro-incisions.
  Arms: FLEX Vessel Prep System followed with PTA (TEST arm)
Device: Angioplasty — The brand and type of PTA balloon(s) used will be at the discretion of the treating physician and used according to its Instructions for Use (IFU). PTA balloons consist of an over-the-wire catheter with a balloon fixed at the distal tip. Within the lesion the balloon is inflated to a pressure that allows full effacement.
  Arms: PTA only (CONTROL arm)

SUMMARY:
A prospective, multi-center, randomized observational post-market study evaluating the FLEX Vessel Prep device plus percutaneous angioplasty (PTA) vs PTA alone for the treatment of obstructive lesions in the native arteriovenous dialysis fistulae.

DETAILED DESCRIPTION:
This is a prospective randomized (1:1) post-market observational study evaluating the FLEX Vessel Prep System followed with PTA vs PTA alone for the treatment of de novo or non-stented restenotic obstructive lesions up to 100 mm in length located in the arteriovenous dialysis fistulae in an upper extremity.

The objective is to evaluate and compare the serious adverse event rate at 30 days and primary patency at 6 months when using FLEX Vessel Prep System prior to PTA vs. PTA alone for treatment of obstructive lesion of native arteriovenous fistulae in the upper extremity.

Enrollment will continue until complete data sets are collected for up to 75 subjects from up to 7 sites in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥21 years of age.
2. Patient has a life expectancy of ≥12 months.
3. Patient has a native AV fistula created ≥ 60 days prior to the index procedure.
4. The target AV fistula has undergone successful dialysis for at least 8 of 12 sessions during a four-week period.
5. Patient has a de novo and/or non-stented restenotic lesion located between approximately 2 cm proximal to the arteriovenous anastomosis and axillosubclavian junction with ≥50% stenosis.
6. Patient has a target lesion (which may include a tandem lesion) that is ≤ 100 mm in length (by visual estimate).

   Note: Tandem lesions may be enrolled provided they meet all of the following criteria:
   * Separated by a gap of ≤ 30mm (3 cm).
   * Total combined lesion length, including 30 mm gap, ≤ 100 mm.
   * Able to be treated as a single lesion.
7. Patient has a target vessel diameter of 4.0 - 12.0 mm (by visual estimate)
8. Patient underwent successful crossing of the target lesion with the guidewire.
9. Patient provides written informed consent prior to enrollment in the study.
10. Patient is willing to comply with all follow-up evaluations at specified times.

Exclusion Criteria:

1. Patient is pregnant or breastfeeding.
2. Patient is receiving immunosuppressive therapy.
3. Patient has undergone prior intervention of access site within 30 days of index procedure.
4. Patient with anticipated conversion to peritoneal dialysis.
5. Patient has an infected AV access or systemic infection.
6. Patient has planned surgical revision of access site.
7. Patient with secondary non-target lesion requiring treatment within 30 days post index procedure.
8. Patient with hemodynamically significant central venous stenoses that cannot be successfully treated prior to treatment of the target lesion.
9. Patient with target AVF or access circuit which previously had thrombectomy within last 30 days.
10. Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the delivery system.
11. Patient with target lesion located central to the axillosubclavian junction.
12. Patient has significant arterial inflow lesion requiring treatment more than 2 cm upstream from the anastomosis in the AV access.
13. Patient has presence of pseudoaneurysm or aneurysm requiring surgical revision at the target lesion site.
14. Patient with known contraindication, including allergic reaction, or sensitivity to contrast material that cannot be adequately pre-treated.
15. Patient who cannot receive recommended antiplatelet and/or anticoagulant therapy.
16. Patient with clinically significant Steal Syndrome requiring treatment.
17. Patient is enrolled in another investigational drug, device, or biologic study and has not completed the primary endpoint or was previously enrolled in this study.
18. Patient has a co-morbid condition that, in the judgment of the Investigator, may cause him/her to be non-compliant with the protocol or confound the data interpretation.
19. Patient has AV fistula created via endovascular technique.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - AKDHC Medical Research Services, Phoenix, Arizona
  - Open Access Vascular Access, Miami, Florida
  - Minneapolis Vascular Surgery Center, New Brighton, Minnesota
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - North Carolina Nephrology, Raleigh, North Carolina
  - Dialysis Access Institute, Orangeburg, South Carolina
  - Dallas Nephrology Associates, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLEX Vessel Prep System Followed With PTA (TEST Arm) | PTA Only (CONTROL Arm)
Started | 38 | 37
Completed | 38 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLEX Vessel Prep System Followed With PTA (TEST Arm) | PTA Only (CONTROL Arm) | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 19 | 17 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 28 | 23 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 35 | 31 | 66
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 21 | 46
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75
Weight [Mean (Full Range); unit: pounds] | 184 [102 to 300] | 171 [116 to 235] | 177 [102 to 300]

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Serious Adverse Event Rate
Description: Defined as the Serious Adverse Event (SAE) rate involving the AV access circuit through 30 days post- procedure.
Time Frame: 30 Days
Measure: Number; unit: percentage of patients
Arm/Group | FLEX Vessel Prep System Followed With PTA (TEST Arm) | PTA Only (CONTROL Arm)
Number analyzed (Participants) | 38 | 37
percentage of patients | 0 | 2.7

ADVERSE EVENTS:
Time Frame: 30 days for primary endpoint
Arm/Group | FLEX Vessel Prep System Followed With PTA (TEST Arm) | PTA Only (CONTROL Arm)
All-Cause Mortality (participants affected / at risk) | 2/38 | 3/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLEX Vessel Prep System Followed With PTA (TEST Arm) (N=38) | PTA Only (CONTROL Arm) (N=37)
Aneurysm of upper arm (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT05034939/Prot_SAP_000.pdf